CLINICAL TRIAL: NCT06177652
Title: Comparison of Thoracal Paravertebral Block and Serratus Plan Block in Pain Management After Thoracotomy
Brief Title: Postoperative Analgesis for Pain Management After Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nur Nazire Yucal, Doctor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: KAEK/10.bI.02
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain; Analgesia
Keywords: Regional Anesthesia; Paravertebral Block; Serratus Plane Block; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single(Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral Block (Active Comparator): Ultrasound (US) -guided paravertebral block (PVB) with 20 ml 0.5 % bupivacaine will performe preoperatively to all patients in the PVB group.
  Interventions: Other: Paravertebral Block
- Serratus Plane Block (Active Comparator): Ultrasound (US) -guided serratus plane block (SPB) with 20 ml 0.5 % bupivacaine will performe preoperatively to all patients in the SPB group.
  Interventions: Other: Serratus Plane Block

INTERVENTIONS:
Other: Paravertebral Block — Ultrasound (US) -guided paravertebral block (PVB) with 20 ml 0.5 % bupivacaine will performe preoperatively to all patients in the PVB group.
  Arms: Paravertebral Block
Other: Serratus Plane Block — Ultrasound (US) -guided serratus plane block (SPB) with 20 ml 0.5 % bupivacaine will performe preoperatively to all patients in the SPB group.
  Arms: Serratus Plane Block

SUMMARY:
Thoracotomy is among the most painful surgical procedures and can cause severe pain. Postoperative pain causes many complications. Therefore, pain management is important in patients undergoing thoracotomy. For this purpose, systemic analgesics are used along with ultrasound-guided nerve blocks in thoracotomy pain. The effectiveness of thoracic paravertebral block and serratus plane block in the treatment of post-thoracotomy pain will be evaluated by comparing their effectiveness and complications on postoperative pain. Since the epidural spread of the thoracic paravertebral block is more effective, the effectiveness of postoperative pain relief will be more effective

DETAILED DESCRIPTION:
Thoracotomy is among the most painful surgical procedures and can cause severe pain. This pain causes postoperative complications in patients who have thoracotomy surgery. Uncontrolled pain can cause respiratory and thromboembolic events. Therefore, effective pain management is important in patients undergoing thoracotomy. Investigators aim to compare the analgesic effectiveness and complications of thoracic paravertebral block and serratus anterior plane block in relieving thoracotomy pain, which is one of the most painful surgical procedures. It is aimed to compare the effectiveness and complications of thoracic paravertebral block and serratus plane block in postoperative pain control after thoracotomy. Providing pain control reduces postoperative complications and reduces hospital stay, which increases patient comfort and reduces costs. In this research, postoperative morphine consumption after block applications will be compared, and patients' analgesic needs will be evaluated according to the participants' VAS score. Post-operative 3rd, 6th, 9th, 12th, 24th. Morphine consumption will be evaluated by monitoring the hours. It will be evaluated whether there is a need for additional analgesics. During the operation, the patient's heart rate, blood pressure, saturation and temperature variable values will be closely monitored. Standard monitoring methods will be used when examining these parameters.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 aged patients
* American Society of Anesthesiologists Classification (ASA) I-II-III patients
* patients who scheduled elective thoracic surgery

Exclusion Criteria:

* American Society of Anesthesiologists Classification (ASA) IV-V patients
* patients with coagulopathy
* patient with infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Morphin consumption | during postoperative 24 hour
  Patient in both groups will provide with intravenous patient-controlled analgesia device containing morphine for postoperative analgesia

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | during postoperative 24 hour
  Visual Analogue Scale (VAS) requires the patient to rate their pain on a defined scale.For example , 0-10 where 0 is no pain and 10 is the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Çardaközü, Study Director — Kocaeli University
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University, Kocaeli
  - Nur Nazire Yucal, Kocaeli

IPD SHARING:
Plan to Share IPD: No